CLINICAL TRIAL: NCT01149395
Title: Can Detection of Fragments of Cleaved E-cadherin in Tissue and/or Blood be of Value for Identifying and Monitoring Patients With PPI-responsive Heartburn?
Brief Title: Can E-cadherin Found in Tissue/Blood be Valuable in Identifying & Monitoring Patients With Post-proton Pump Inhibitor (PPI)-Responsive Heartburn
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10-0417
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Heartburn; Gastroesophageal Reflux Disease
Keywords: Heartburn; Gastroesophageal Reflux Disease
MeSH Terms: conditions — Heartburn; Gastroesophageal Reflux | interventions — Dexlansoprazole; Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexlansoprazole (Experimental)
  Interventions: Drug: Dexlansoprazole

INTERVENTIONS:
Drug: Dexlansoprazole — Dosage: 30 mg once per day for 4 weeks by mouth
  Other Names: Kapidex

SUMMARY:
The purpose of this research study is to determine in heartburn patients with nonerosive disease if detecting the presence of a fragment of the protein e-cadherin in esophageal epithelium or the amount of fragments of e-cadherin in blood can be used to monitor healing of esophagitis treated with a proton pump inhibitor (PPI). The hypothesis is that the presence of fragments of e-cadherin in esophageal epithelium or the amount of fragments of e-cadherin in blood can you useful as a biomarker for the healing of esophagitis in patients successfully treated with a PPI.

DETAILED DESCRIPTION:
The symptom of heartburn was once a reliable indicator of gastroesophageal reflux disease (GERD) and as such patients would predictably respond to acid inhibition. In the post-proton pump inhibitor (PPI) world, neither of these statements is true since many patients presenting with heartburn have symptoms mediated by mechanisms unrelated to esophageal luminal acidity, e.g. functional disease, visceral hypersensitivity or activation of esophageal stretch receptors. Consequently these subjects fail to respond to PPIs[1-3]. Since PPI-responsive and PPI-refractory patients with heartburn are indistinguishable by history, it is difficult to determine which PPI-unresponsive subjects may respond to higher doses of a PPI. Additionally, when subjects do respond to PPI therapy, symptom response may not correlate with lesion healing, making a systemic marker of healing highly desirable. Lesion healing is particularly problematic since the histopathologic lesion that correlates best with heartburn is the presence of dilated intercellular spaces (DIS) within esophageal epithelium, which cannot be detected by with standard endoscopy, and is most reliably demonstrable by performing transmission electron microscopy[4-7]. Consequently, it would be desirable to have an objective marker of acid-mediated injury to esophageal epithelium that could identify those with PPI-responsive heartburn and determine healing of acid-damaged epithelium non-invasively.

DIS in esophageal epithelium has been established as an early histopathologic feature of gastroesophageal reflux disease (GERD). This electron microscopic lesion is present in both erosive and nonerosive forms of GERD and results from acid damage to the intercellular junctional complex that controls paracellular permeability within esophageal epithelium[8]. Further, it is known that treatment with PPIs results in resolution of DIS along with that of heartburn in patients with both erosive and nonerosive types of GERD[9]. E-cadherin is a protein which forms the intercellular adhesive bridge of the zonula adherens (ZA)[10]; and the ZA plays an integral role in maintaining the integrity of the tight junction between cells such that loss of adhesion between bridging molecules of e-cadherin results in loss of barrier function and increased paracellular permeability[11,12]. Therefore, under conditions where an acidic refluxate is present within the esophageal lumen, a 'leaky' junctional barrier promotes excessive entry of hydrogen ions into and so acidification of the intercellular space, which in turn triggers heartburn by activation of acid-sensitive neurons within the mucosa[13].

Recently, my lab has found that DIS in non-erosive acid-damage to (rabbit) esophageal epithelium is associated on Western blots with cleavage of the intercellular portion of e-cadherin and that this cleavage occurs by acid activation of an endogenous proteolytic process (unpublished observations). Moreover, this same phenomenon on Western blots is replicated in human esophagus of patients with GERD, i.e. endoscopic biopsies of esophageal epithelium reveal cleavage of e-cadherin in those with both erosive and non-erosive forms of GERD but is not present within the esophageal epithelium of healthy subjects or subjects without signs or symptoms of esophageal disease[14] - see Fig 4 of attached poster presentation. Specifically, cleavage of e-cadherin in GERD patients leaves behind within the esophageal epithelium a cytoplasmic 'C-terminal fragment (CTF)' of the molecule and this CTF is readily detected on Western blot. Interestingly, the size of the CTF is consistent, as in the rabbit model, with cleavage of e-cadherin by an endogenous matrix metalloprotease. Also noteworthy is that the other cleaved extracellular component of e-cadherin is an 'N-terminal fragment (NTF)' and this fragment is absorbed into the blood stream resulting in higher serum levels of NTFs of e-cadherin than healthy subjects as detectable using a commercial ELISA assay[14] - see Fig. 6 of attached poster presentation. Since CTFs on Western blot of endoscopic biopsies and elevated NTFs of e-cadherin by ELISA in serum are a reflection of acid-injured esophageal epithelium, this suggests the tantalizing possibility of a sensitive, minimally invasive (serum) test for esophageal mucosal damage in the GERD subject. We hypothesize that determination of either of the cleaved fragments of e-cadherin (serum or tissue-based) can discriminate between patients with acid-mediated heartburn who are likely to be PPI-responsive and those whose heartburn symptoms are not mediated by acid and so are PPI-refractory.

The hypothesis will be tested by determining the presence or absence of CTFs of e-cadherin on esophageal biopsy and by measuring the level of NTFs of e-cadherin in serum of endoscopy-negative patients with heartburn and correlating the findings with the patient's (heartburn) response to Kapidex 30 mg for 4 weeks. Based on effective heartburn control on Kapidex or lack thereof, patients will be classified as having PPI-responsive or PPI-refractory disease, respectively, and these classifications correlated with presence or absence of CTFs on pretreatment biopsy and pretreatment serum level of NTFs of e-cadherin. Also, after 4 weeks of Kapidex, repeat serum specimens for NTFs are obtained from all treated patients to determine, as a marker of healing, whether the serum level of NTFs post-treatment are significantly lower than pretreatment serum level of NTFs in those that have PPI-responsive heartburn but not in those that have PPI-refractory heartburn.

The results of this study are expected to show that patients with PPI-responsive heartburn have CTFs of e-cadherin in tissue and higher levels of NTFs of e-cadherin in serum at baseline, and that these levels decrease after successful PPI therapy. In contrast, because symptoms in PPI-refractory subjects are not acid-mediated, these subjects are expected to lack CTFs in tissue and to have lower levels of NTFs in serum at baseline compared to PPI-responsive patients, and these levels will remain unchanged after PPI therapy. Consequently, such findings would establish detection of cleaved fragments of e-cadherin in tissue and blood as useful biomarkers of disease that can identify those with heartburn that are responsive to standard doses of Kapidex. The results are also expected to show that patients with PPI-responsive heartburn, but not those with PPI-refractory heartburn, have a significant decline in the level of NTFs in serum post-treatment and that this lower level of NTFs is expected to fall within the range of controls. Consequently, such findings would establish that detection of serum NTFs before and after treatment can be useful as a biomarker of (microscopic) lesion healing in those with PPI-responsive heartburn. Such findings might help select sub-groups appropriate for more intensive (higher dose) or long term PPI therapy.

ELIGIBILITY:
Inclusion Criteria: (all responses must be Yes)

* Between 18 and 75 years of age
* Male or non-pregnant, non-lactating female
* Willing and able to undergo endoscopy with biopsies and a blood draw
* Willing and able to discontinue use of PPIs for at least 1 month prior to the study start date
* Endoscopy-negative heartburn of moderate severity at least 3 times-a-week for 3 months

Exclusion Criteria:(all responses must be No)

* History of:

  * Barrett's Esophagus
  * Erosive Esophagus
  * Zollinger Ellison syndrome
  * bleeding disorder
  * upper gastrointestinal bleeding or malignancy
  * esophageal motor disorder
  * esophageal stricture
  * esophageal varices
* Had the following surgeries:

  * organ transplant
  * gastric or esophageal surgery for the treatment of: Esophageal Cancer, Achalasia, Gastroesophageal Reflux Disease (GERD); i.e. Nissen Fundoplication
* Have any of the following:

  * Current malabsorption
  * inflammatory bowel disease
  * severe heart-lung-liver or renal cerebrovascular disease
  * known hypersensitivity to PPIs
* Currently taking any of the following medications:

  * Quinidine
  * quinine
  * benzodiazepines
  * antineoplastic agents
  * dilantin
  * warfarin
  * non-steroidal anti-inflammatory drugs
  * narcotics
  * prostaglandins
  * salicylates (except baby aspirin for cardiovascular protection)
  * H2-receptor antagonists
  * PPIs other than study agent
  * steroids
  * promotability drugs
  * sucralfate
  * KCl
  * anti-tuberculosis medication
  * oral biphosphonates
  * drugs requiring acid for absorption (iron, ampicillin, digoxin and ketoconazole)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Dexlansoprazole | 4 weeks
  Primary outcome measure: To determine whether detection of cleaved fragments of e-cadherin in esophageal biopsies and in serum can discriminate between nonerosive patients with PPI-responsive and PPI-refractory heartburn.

SECONDARY OUTCOMES:
Dexlansoprazole | 4 weeks
  To determine whether serum levels of N-terminal fragments of e-cadherin can be useful to monitor esophageal healing in patients with nonerosive PPI-responsive heartburn.

CONTACTS AND LOCATIONS:
Overall Officials: Roy C Orlando, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States